CLINICAL TRIAL: NCT06377267
Title: Non-Randomized, Open-Label, Prospective Phase II Trial to Better Characterize the Status of HRD Leading to a Benefit From Olaparib in Combination With Bevacizumab in Patients With Advanced FIGO Stage III-IV High Grade Serous or Endometrioid Ovarian, Fallopian Tube, or Peritoneal Cancer After Standard First-Line Treatment
Brief Title: Status of HRD That Lead to a Benefit From Olaparib in Combination With Bevacizumab (STROBE Trial)
Acronym: STROBE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-20-21103
Record Dates: First submitted 2024-04-10; First posted 2024-04-22 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Cancer
Keywords: HRD status
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRD positive arm (Experimental): Patient with harboring HRD tumor, that will receive olaparib in combination with bevacizumab
  Interventions: Drug: Bevacizumab; Drug: Olaparib
- HRD negative arm (Other): Control group receiving bevacizumab alone as standard of care.Patient with non harboring HRD tumor, that will receive bevacizumab
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab dosing is at 15 mg/kg every 3 weeks as an intravenous infusion.
Drug: Olaparib — Olaparib dosing is oral at 300 mg twice daily
  Arms: HRD positive arm

SUMMARY:
Background:

The study aims to address the challenge of accurately identifying patients with ovarian cancer who would benefit from poly-ADP ribose inhibitors (PARPi) as first-line maintenance therapy. While BRCA1/2-mutated epithelial ovarian cancer (EOC) patients have shown significant benefits from PARPi treatment, the efficacy in homologous recombination deficient (HRD) patients remains inconclusive. Current assays used to estimate HR status do not effectively differentiate between patients who benefit most from PARPi and those who do not, making it inefficient to treat all patients. There is a need for a more accurate HR status testing method to optimize PARPi benefit. This study aims to assess the performance of the VHIO-CARD-300 test in determining HR status compared to SOPHiA DDM™ Dx HRD Solution.

Summary:

The study is a prospective, non-randomized trial designed to evaluate the concordance of the VHIO-CARD-300 test in establishing HR status compared to SOPHiA DDM™ Dx HRD Solution. Additionally, it aims to assess the association between HRD status determined by the VHIO-CARD-300 test and treatment efficacy. Patients with advanced FIGO stage III-IV high grade serous or endometrioid ovarian, fallopian tube, or peritoneal cancer will be invited to participate. Those eligible will undergo testing with both VHIO-CARD-300 and SOPHiA DDM™ Dx HRD Solution. Patients classified as HRD positive will receive olaparib in combination with bevacizumab, while others will receive bevacizumab alone. Treatment will be administered according to approved doses, with follow-up evaluations conducted until RECIST progression.

DETAILED DESCRIPTION:
This non-randomized, open-label phase II trial seeks to enhance our understanding of HRD status in patients with advanced ovarian, fallopian tube, or peritoneal cancer. Following standard first-line treatment, participants will be assessed for HRD status using the VHIO-CARD-300 test and SOPHiA DDM™ Dx HRD Solution. Those identified as HRD-positive will receive olaparib in combination with bevacizumab, while others will receive bevacizumab alone as per standard care. The study aims to determine the concordance between the two HRD tests, evaluate the efficacy of the olaparib-bevacizumab combination, and assess safety and tolerability. Efficacy outcomes will be evaluated using RECIST criteria, with a minimum follow-up of 30 months post-enrollment. Secondary objectives include examining treatment accuracy, association with efficacy outcomes, and analyzing discrepant cases. Overall, this trial aims to provide valuable insights into personalized treatment approaches for patients with advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with newly diagnosed high- grade serous or endometrioid Ovarian cancer, primary peritoneal cancer and/or fallopian-tube cancer. I-3-3 At an advanced stage: FIGO stage IIIB, IIIC, or IV of the 1988 FIGO classification (see appendix 1).
2. Patient who has completed prior to enrollment first line platinum-taxane chemotherapy:

   1. Platinum-taxane based regimen must have consisted of
   2. minimum of 6 treatment cycles and a maximum of 8. However, if platinum-based therapy must be discontinued early as a result of non-hematological toxicityspecificallyrelated to the platinum regimen, (i.e. neurotoxicity, hypersensitivity etc.), patient must have received a minimum of 4 cycles of the platinum regimen.
   3. Patient must have received prior to enrollment a minimum of 3 cycles of bevacizumab in combination with the 3 last cycles of platinum-based chemotherapy. Only in case of interval debulking surgery, it is allowed to realize only 2 cycles of bevacizumab in combination with the last 3 cycles of platinum-based chemotherapy.
3. Patient must be prior to enrollment without evidence of disease (NED) or in complete response (CR) or partial response (PR) from the first line treatment. There should be no clinical evidence of disease progression (physical exam, imagery, CA 125) throughout he first line treatment and prior to study enrollment.
4. Patient must be randomized at least 4 weeks and no more than 8 weeks after her last dose of chemotherapy (last dose is the day of the last infusion) and all major toxicities from theprevious chemotherapy must have resolved to CTCAE grade 1 or better (except alopecia and peripheral neuropathy).
5. Patient must have normal organ and bone marrow function:
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (see appendix 3)
7. Formalin fixed, paraffin embedded (FFPE) tumor sample from the primary cancer must be available for central BRCA testing and test result must be available for stratification.

Exclusion Criteria:

1. Non-epithelial origin of the ovary, the fallopian tube or the peritoneum (i.e. germ cell tumors).
2. Ovarian tumors of low malignant potential (e.g. borderline tumors) or mucinous carcinoma.
3. Other malignancy within the last 5 years except:
4. Patient with myelodysplastic syndrome/acute myeloid leukemia history.
5. Major surgery within 4 weeks of starting study treatment and patient must have recovered from any effects of any major surgery.
6. Any previous treatment with PARP inhibitor, including olaparib.
7. Concomitant use of known potent CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir.
8. Prior history of hypertensive crisis (CTC-AE grade 4) or hypertensive encephalopathy.
9. Clinically significant (e.g. active) cardiovascular disease, including:

   1. Myocardial infarction or unstable angina within ≤ 6 months of enrollment,
   2. New York Heart Association (NYHA) ≥ grade 2 congestive heart failure (CHF) (see appendix 5).
   3. Poorly controlled cardiac arrhythmia despite medication (patient with rate controlled atrial fibrillation are eligible), or any clinically significant abnormal finding on resting ECG,
   4. Peripheral vascular disease grade ≥ 3 (e.g. symptomatic and interfering with activities of daily living [ADL] requiring repair or revision)
10. Previous Cerebro-Vascular Accident (CVA), Transient Ischemic Attack (TIA) or Sub-Arachnoids Hemorrhage (SAH) within 6 months prior to enrollment.
11. History or evidence of hemorrhagic disorders within 6 months prior to enrollment.
12. History or clinical suspicion of brain metastases or spinal cord compression.
13. Significant traumatic injury during 4 weeks prior to enrollment.
14. Non-healing wound, active ulcer or bone fracture.
15. History of VEGF therapy related abdominal fistula or gastrointestinal perforation or active gastrointestinal bleeding within 6 months prior to the first study treatment.
16. Current, clinically relevant bowel obstruction, including sub-occlusive disease, related to underlying disease.
17. Patient with evidence of abdominal free air not explained by paracentesis or recent surgical procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Concordance in HRD status identification between VHIO-CARD-300 test and SOPHiA DDM™ Dx HRD Solution | Through study completion, an average of 1.5 years
  The primary outcome measure description would outline the method used to evaluate the agreement in HRD status identification between the VHIO-CARD-300 test and SOPHiA DDM™ Dx HRD Solution. This would include details on how HRD status is determined and compared between the two tests, along with any statistical analyses employed to measure the level of agreement.

SECONDARY OUTCOMES:
Performance Assessment of VHIO-CARD-300 Test for HR Status Identification | Through study completion, an average of 1.5 years
  This secondary outcome measure focuses on evaluating the performance of the VHIO-CARD-300 test as a diagnostic tool for identifying HR status. The assessment will include determining the sensitivity, specificity, and predictive positive and negative values of the VHIO-CARD-300 test, with the SOPHiA DDM™ Dx HRD Solution serving as the reference standard.
Association Between VHIO-CARD-300 Test Groups and Efficacy Outcomes(i.e., HRD positive and HRD negative) and efficacy outcomes. | Through study completion, an average of 1.5 years
  To assess the relationship between the HRD positive and HRD negative groups identified by the VHIO-CARD-300 test and treatment efficacy outcomes.
Analysis of Progression-Free Survival (PFS) and Overall Survival (OS) in Discrepant HRD Cases | Through study completion, an average of 1.5 years
  This outcome measure aims to assess the efficacy outcomes in cases where there is a discrepancy between the results obtained from the VHIO-CARD-300 test and the SOPHiA DDM™ Dx HRD Solution. Specifically, it focuses on cases where a patient is classified as HRD positive by one test but HRD negative by the other, and vice versa. The primary efficacy endpoints, progression-free survival (PFS) and overall survival (OS), will be analyzed in these discrepant cases to evaluate the impact of the discordant results on clinical outcomes
Safety and Tolerability of Olaparib Plus Bevacizumab | Through study completion, an average of 1.5 years
  Assessment of adverse events (AEs) graded by the National Cancer Institute (NCI) CTCAE v5.0, serious adverse events (SAEs), abnormal vital signs, abnormal ECG results, and evaluation of laboratory parameters
To evaluate the failure rate for the VHIOCARD-300 test and SOPHiA DD Dx HRD Solution. | Through study completion, an average of 1.5 years
  Percentage of inconclusive results will be estimated for each test

CONTACTS AND LOCATIONS:
Overall Officials: Ana Oaknin, Principal Investigator — Vall d'Hebron Institute of Oncology
Locations (1):
- Vall d'Hebron Institute of Oncology, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No